CLINICAL TRIAL: NCT04511000
Title: A Randomized, Open-label, Parallel, Multi-Center Phase IV Study to Compare of the Efficacy and Safety of Lipilou 20 mg and Lipilou 10 mg in High-risk Patients With Hypercholesterolemia(PEARL Study)
Brief Title: Clinical Trial to to Compare of the Efficacy and Safety of Lipilou® 20 mg and Lipilou® 10 mg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 124HL17003
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Lipilou®(generic atorvastatin drug) 20 mg
- Comparator group (Active Comparator)
  Interventions: Drug: Lipilou®(generic atorvastatin drug) 10 mg

INTERVENTIONS:
Drug: Lipilou®(generic atorvastatin drug) 20 mg — Patients assigned to experimental group are treated with Lipilou® 20 mg
  Arms: Experimental group
Drug: Lipilou®(generic atorvastatin drug) 10 mg — Patients assigned to comparator group are treated with Lipilou® 10 mg
  Arms: Comparator group

SUMMARY:
This study was designed to compare the mean percent change of LDL-C between Lipilou® 10mg and 20mg group after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had hypercholesterolemia with high risk, according to the 2015 Korean guidelines for managing dyslipidemia.

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus, uncontrolled hypertension, thyroid dysfunction.
* Patients who are legally unable to participate in clinical trials or who are unable to participate in clinical trials based on investigator's decision.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Change rate in LDL-C | 12 weeks of treatment
  compare experimental group with comparator group

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Korea University Ansan Hospital, Ansan
  - Sejong General Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Inje University Ilsan Paik Hospital, Goyang
  - Myongji Hospital, Goyang
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan